CLINICAL TRIAL: NCT01458535
Title: An Open-Label, Sequential Arm, Multicenter Study to Evaluate the Antiviral Activity, Safety and Pharmacokinetics of ABT-450 With Ritonavir (ABT-450/r) Dosed in Combination With ABT-267 With and Without Ribavirin (RBV) in Treatment-Naïve Subjects With Genotype 1, 2 or 3 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Study to Evaluate Paritaprevir With Ritonavir (ABT-450/r) When Given Together With Ombitasvir and With and Without Ribavirin (RBV) in Treatment-Naïve Participants With Genotype 1, 2 or 3 Chronic Hepatitis C Virus (HCV)
Acronym: Navigator
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-998
Record Dates: First submitted 2011-09-23; First posted 2011-10-25 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C Virus
Keywords: Genotype 1; Genotype 2; Genotype 3; Hepatitis C Virus; ABT-450/r; Ribavirin; ABT-267; Ombitasvir; Paritaprevir
MeSH Terms: conditions — Hepatitis C | interventions — paritaprevir; ombitasvir; Ribavirin; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- ABT-450/r and ABT-267 plus RBV in genotype 1 participants (Experimental): ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD plus weight-based ribavirin (RBV) divided twice daily (BID) in treatment-naïve participants with HCV genotype 1 infection.
  Interventions: Drug: ABT-450; Drug: ABT-267; Drug: ribavirin; Drug: ritonavir
- ABT-450/r and ABT-267 plus RBV in genotype 2 participants (Experimental): ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD plus weight-based ribavirin (RBV) divided BID in treatment-naïve participants with HCV genotype 2 infection.
  Interventions: Drug: ABT-450; Drug: ABT-267; Drug: ribavirin; Drug: ritonavir
- ABT-450/r and ABT-267 plus RBV in genotype 3 participants (Experimental): ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD plus weight-based ribavirin (RBV) divided BID in treatment-naïve participants with HCV genotype 3 infection.
  Interventions: Drug: ABT-450; Drug: ABT-267; Drug: ribavirin; Drug: ritonavir
- ABT-450/r and ABT-267 in genotype 1 participants (Experimental): ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD in treatment-naïve participants with HCV genotype 1 infection.
  Interventions: Drug: ABT-450; Drug: ABT-267; Drug: ritonavir
- ABT-450/r and ABT-267 in genotype 2 participants (Experimental): ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD in treatment-naïve participants with HCV genotype 2 infection.
  Interventions: Drug: ABT-450; Drug: ABT-267; Drug: ritonavir
- ABT-450/r and ABT-267 in genotype 3 participants (Experimental): ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD in treatment-naïve participants with HCV genotype 3 infection.
  Interventions: Drug: ABT-450; Drug: ABT-267; Drug: ritonavir

INTERVENTIONS:
Drug: ABT-450 — tablets
  Other Names: paritaprevir
Drug: ABT-267 — tablets
  Other Names: ombitasvir
Drug: ribavirin — tablets
  Arms: ABT-450/r and ABT-267 plus RBV in genotype 1 participants; ABT-450/r and ABT-267 plus RBV in genotype 2 participants; ABT-450/r and ABT-267 plus RBV in genotype 3 participants
Drug: ritonavir — capsules
  Other Names: Norvir

SUMMARY:
The purpose of this study was to evaluate the efficacy, safety and pharmacokinetics of ABT-450/r when given together with ABT-267 and with and without RBV in treatment-naïve participants with genotype 1, 2 or 3 chronic HCV infection.

DETAILED DESCRIPTION:
This was a 2 sequential arm, combination treatment study where each arm contained 3 cohorts: one each for HCV genotype 1, 2, and 3. The study consisted of 2 phases, a treatment phase and a post-treatment phase. The treatment phase was designed to explore the antiviral activity, safety and pharmacokinetics of ABT-450/r dosed in combination with ABT-267 with and without RBV for up to 12 weeks. The post-treatment phase was designed to monitor and evaluate Sustained Virologic Response (SVR) 12, SVR 24, and the evolution and persistence of viral resistance to ABT-267 and ABT-450 in HCV genotype 1-, 2-, and 3-infected participants who have been exposed to ABT-267 and ABT-450/r. Arms 1 and 2 were enrolled sequentially.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had a body mass index 18 to < 35 kg/m^2.
* Females were either postmenopausal for at least 2 years, surgically sterile, or willing to use at least 2 effective forms of birth control.
* Males must have been surgically sterile or agreed to use at least 2 effective forms of birth control throughout the course of the study.
* Participants were in a condition of general good health, other than the HCV infection.
* Participants had a chronic HCV genotype 1, 2, or 3 infection for at least 6 months, a plasma HCV RNA > 50,000 IU/mL, and FibroTest score <= 0.72 and aspartate aminotransferase (AST) to platelet ratio index <= 2, Fibroscan® result of < 9.6 kilopascal (kPa), or absence of cirrhosis based on a liver biopsy.

Exclusion Criteria:

* Positive drug screen
* Previous use of anti-HCV agents
* History of cardiac disease
* History of uncontrolled diabetes or diabetes requiring insulin
* Abnormal laboratory results
* Females who were pregnant or planned to become pregnant within 6 months after their last dose of study drug/RBV or were breastfeeding; males whose partners were pregnant or would become pregnant within 6 months after their last dose of study drug/RBV
* Positive test result for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus (HIV) antibody (Ab). Negative HIV status was to be confirmed at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Campbell, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants: ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD plus weight-based ribavirin (RBV) divided twice daily (BID) in treatment-naïve genotype 1 participants.
- ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants: ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD plus weight-based ribavirin (RBV) divided BID in treatment-naïve genotype 2 participants.
- ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants: ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD plus weight-based ribavirin (RBV) divided BID in treatment-naïve genotype 3 participants.
- ABT-450/r and ABT-267 in Genotype 1 Participants: ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD in treatment-naïve genotype 1 participants.
- ABT-450/r and ABT-267 in Genotype 2 Participants: ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD in treatment-naïve genotype 2 participants.
- ABT-450/r and ABT-267 in Genotype 3 Participants: ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD in treatment-naïve genotype 3 participants.
Period: Overall Study
Arm/Group | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants | ABT-450/r and ABT-267 in Genotype 1 Participants | ABT-450/r and ABT-267 in Genotype 2 Participants | ABT-450/r and ABT-267 in Genotype 3 Participants
Started | 10 | 10 | 10 | 10 | 10 | 11
Completed | 10 | 8 | 8 | 6 | 6 | 7
Not Completed | 0 | 2 | 2 | 4 | 4 | 4
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0 | 3 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants: ABT-450/r (200/100 mg) once daily (QD) and ABT-267 (25 mg) QD plus weight-based ribavirin (RBV) divided BID in treatment-naïve genotype 1 participants.
- Total: Total of all reporting groups
Arm/Group | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants | ABT-450/r and ABT-267 in Genotype 1 Participants | ABT-450/r and ABT-267 in Genotype 2 Participants | ABT-450/r and ABT-267 in Genotype 3 Participants | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (12.19) | 51.1 (8.25) | 40.3 (13.10) | 45.9 (7.03) | 54.9 (10.85) | 48.7 (8.91) | 47.6 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 3 | 7 | 3 | 4 | 27
  Male | 2 | 8 | 7 | 3 | 7 | 7 | 34
HCV Genotype/ Subtype [Number; unit: participants]
  1A | 8 | 0 | 0 | 8 | 0 | 0 | 16
  1B | 2 | 0 | 0 | 2 | 0 | 0 | 4
  2A | 0 | 2 | 0 | 0 | 2 | 0 | 4
  2B | 0 | 8 | 0 | 0 | 8 | 0 | 16
  3A | 0 | 0 | 10 | 0 | 0 | 11 | 21
  3B | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interleukin 28B (IL28B) [Number; unit: participants]
  CC | 1 | 2 | 2 | 4 | 4 | 3 | 16
  CT | 7 | 4 | 7 | 4 | 5 | 7 | 34
  TT | 2 | 4 | 1 | 2 | 1 | 1 | 11
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Suppressed Below the Lower Limit of Quantitation (LLOQ) From Week 4 Through Week 12 [(Extended Rapid Virologic Response (eRVR)]
Description: Analysis of the percentage of participants with hepatitis C virus ribonucleic acid less than the lower limit of quantitation (< 25 IU/mL). Participants with missing data were imputed as failures.
Time Frame: Week 4 through Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants | ABT-450/r and ABT-267 in Genotype 1 Participants | ABT-450/r and ABT-267 in Genotype 2 Participants | ABT-450/r and ABT-267 in Genotype 3 Participants
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11
percentage of participants | 100 | 90.0 | 70.0 | 90.0 | 80.0 | 18.2
Statistical Analysis 1: Comparison: ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants vs ABT-450/r and ABT-267 in Genotype 1 Participants; Test type: Superiority or Other; p = 0.157, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants vs ABT-450/r and ABT-267 in Genotype 2 Participants; Test type: Superiority or Other; p = 0.999, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants vs ABT-450/r and ABT-267 in Genotype 3 Participants; Test type: Superiority or Other; p = 0.045, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks (SVR12) Post-treatment
Description: Sustained Virologic Response 12 (SVR12) is defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (< LLOQ; < 25 IU/mL) 12 weeks after the last dose of study drug. Participants with missing data were imputed as failures.
Time Frame: Post-treatment Day 1 to Post-treatment Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants | ABT-450/r and ABT-267 in Genotype 1 Participants | ABT-450/r and ABT-267 in Genotype 2 Participants | ABT-450/r and ABT-267 in Genotype 3 Participants
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11
percentage of participants | 100 | 80.0 | 50.0 | 60.0 | 60.0 | 9.1

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks (SVR24) Post-Treatment
Description: Sustained Virologic Response 24 (SVR24) is defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ; < 25 IU/mL) 24 weeks after the last dose of study drug. Participants with missing data were imputed as failures.
Time Frame: Post-treatment Day 1 to Post-treatment Week 24
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants | ABT-450/r and ABT-267 in Genotype 1 Participants | ABT-450/r and ABT-267 in Genotype 2 Participants | ABT-450/r and ABT-267 in Genotype 3 Participants
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11
percentage of participants | 100 | 80.0 | 40.0 | 60.0 | 60.0 | 9.1

4. Secondary Outcome: Percentage of Participants With Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) < 1000 International Units Per Milliliter (IU/mL)
Description: Analysis of participants with HCV RNA levels below 1000 IU/mL at Week 2. Participants with missing data were imputed as failures.
Time Frame: Week 2
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants | ABT-450/r and ABT-267 in Genotype 1 Participants | ABT-450/r and ABT-267 in Genotype 2 Participants | ABT-450/r and ABT-267 in Genotype 3 Participants
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100

5. Secondary Outcome: Percentage of Participants With Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Below the Lower Limit of Quantitation (LLOQ) at Week 4 Rapid Virologic Response (RVR)
Description: Analysis of percentage of participants with hepatitis C virus ribonucleic acid less than the lower limit of quantitation (< 25 IU/mL). Participants with missing data were imputed as failures.
Time Frame: Week 4
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants | ABT-450/r and ABT-267 in Genotype 1 Participants | ABT-450/r and ABT-267 in Genotype 2 Participants | ABT-450/r and ABT-267 in Genotype 3 Participants
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11
percentage of participants | 100 | 100 | 90.0 | 100 | 90.0 | 27.3

6. Secondary Outcome: Percentage of Participants With Virologic Failure During Treatment
Description: Virologic failure during treatment is defined as a participant meeting any virologic stopping criteria, including 1) rebound (defined as the first day of 2 consecutive increases of at least 0.5 log10 IU/mL above nadir (local minimum value), or first day of 2 consecutive HCV RNA >= LLOQ for participants who previously achieved HCV RNA < LLOQ) during treatment, 2) participant who fails to suppress (defined as never achieving HCV RNA < LLOQ during treatment).
Time Frame: Day 1 through Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants | ABT-450/r and ABT-267 in Genotype 1 Participants | ABT-450/r and ABT-267 in Genotype 2 Participants | ABT-450/r and ABT-267 in Genotype 3 Participants
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11
percentage of participants
  Participant Rebounds | 0 | 10.0 | 30.0 | 10.0 | 10.0 | 72.7
  Participants who fail to Suppress | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Who Experienced Virologic Relapse Through End of Post Treatment Period (up to 48 Weeks)
Description: Virologic relapse is defined as confirmed hepatitis C virus (HCV) ribonucleic acid (RNA) >= lower limit of quantitation (LLOQ) (2 consecutive measurements >= LLOQ) at any point in the post-treatment period among participants with HCV RNA < LLOQ at the end of treatment. Participants with missing data were imputed as failures.
Time Frame: Post-treatment Day 1 to Post-treatment Week 48
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT) with hepatitis C virus (HCV) ribonucleic acid (RNA) < lower limit of quantitation (LLOQ) at the final treatment visit who completed treatment.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants | ABT-450/r and ABT-267 in Genotype 1 Participants | ABT-450/r and ABT-267 in Genotype 2 Participants | ABT-450/r and ABT-267 in Genotype 3 Participants
Number analyzed (Participants) | 10 | 9 | 7 | 9 | 9 | 2
percentage of participants | 0 | 0 | 28.6 | 22.2 | 22.2 | 50.0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the time of study drug administration to 30 days after last dose of study drug (12 weeks); SAEs were also collected from the time that informed consent was obtained until the end of the study (up to 60 weeks).
Arm/Group | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants | ABT-450/r and ABT-267 in Genotype 1 Participants | ABT-450/r and ABT-267 in Genotype 2 Participants | ABT-450/r and ABT-267 in Genotype 3 Participants
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/10 | 1/10 | 1/10 | 1/11
Other Adverse Events (participants affected / at risk) | 9/10 | 9/10 | 8/10 | 9/10 | 9/10 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants (N=10) | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants (N=10) | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants (N=10) | ABT-450/r and ABT-267 in Genotype 1 Participants (N=10) | ABT-450/r and ABT-267 in Genotype 2 Participants (N=10) | ABT-450/r and ABT-267 in Genotype 3 Participants (N=11)
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
MENINGITIS HERPES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
TRAUMATIC LIVER INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r and ABT-267 Plus RBV in Genotype 1 Participants (N=10) | ABT-450/r and ABT-267 Plus RBV in Genotype 2 Participants (N=10) | ABT-450/r and ABT-267 Plus RBV in Genotype 3 Participants (N=10) | ABT-450/r and ABT-267 in Genotype 1 Participants (N=10) | ABT-450/r and ABT-267 in Genotype 2 Participants (N=10) | ABT-450/r and ABT-267 in Genotype 3 Participants (N=11)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPERACUSIS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
GROWTH OF EYELASHES (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
VISION BLURRED (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 2 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
ERUCTATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
FAECES PALE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 6 | 3 | 1 | 2 | 2 | 1
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 6 | 3 | 2 | 4 | 3 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
IRRITABILITY (General disorders) | 0 | 1 | 0 | 1 | 2 | 0
MALAISE (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
PAIN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
GROIN INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
KIDNEY INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 1
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
TONGUE ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
URINE OUTPUT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 1 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 1 | 0
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 4 | 2 | 1 | 1 | 1 | 2
LETHARGY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
MIGRAINE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
SINUS HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
AGITATION (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0
PANIC ATTACK (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
BREAST TENDERNESS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
CYSTOCELE (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 2 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
HYPOTENSION (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.